CLINICAL TRIAL: NCT06816550
Title: A Prospective Study of Pattern of Chronic Use of NSAIDS in Patients Admitted to Emergency Department in Alexandria Main University Hospital.
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: 0306890
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-02

CONDITIONS: NSAIDs Administration
Keywords: NSAIDS; chronic use

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients admitted to emergency department in Alexandria Main University Hospital.: patients admitted to emergency department in Alexandria Main University Hospital for detection of patients on chronic use of nonsteroidal anti inflammatory drugs
  Interventions: Other: Doing Interviews with the patients admitted to emergency department to detect whom are on chronic use of nonsteroidal anti inflammatory drugs

INTERVENTIONS:
Other: Doing Interviews with the patients admitted to emergency department to detect whom are on chronic use of nonsteroidal anti inflammatory drugs — detection of patients on chronic use of nonsteroidal anti inflammatory drugs among total patients admitted to emergency department in Alexandria Main University Hospital

SUMMARY:
The goal of this observational study is to assess the pattern of chronic use of nonsteroidal anti inflammatory drugs in patients admitted to emergency department in Alexandria Main University Hospital. The main question it aims to answer is:

What is the prevalence of chronic use of nonsteroidal anti inflammatory drugs among patients admitted to emergency department in Alexandria Main University Hospital?

DETAILED DESCRIPTION:
This is a prospective cross sectional study of pattern of chronic use of NSAIDS in patients admitted to emergency department in Alexandria Main University Hospital.

Three well trained emergency clinical pharmacists will start medication reconciliation process on admission by interviews with the patients or their care givers.

The study aims to assess the pattern of chronic use of NSAIDS and evaluate the patients' knowledge about doses, duration and adverse events and other use precautions .Finally to provide counseling service regarding NSAIDS medical information to patients admitted to emergency department in Alexandria Main University Hospital.

ELIGIBILITY:
Inclusion Criteria: all adults equal or more than 18 years -

Exclusion Criteria:Patients who cannot communicate or have no family members.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to Emergency department in Alexandria main University Hospital during the study period
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
prevelence of chronic use of NSAIDS among total patients admitted to emergency department | two months from 1 March 2025 to 1 May 2025
  (Number of of chronic use of NSAIDS / total patients admitted to emergency department) x 100

SECONDARY OUTCOMES:
Percentage of patients who are already aware about NSAIDS chronic use adverse effects | one month
  Number of patients who are already aware about NSAIDS chronic use adverse effects / total number of patients who are chronic users of NSAIDS x100

OTHER OUTCOMES:
Penrcentage of patients who have taken a counselling session about NSAIDS chronic use adverse effects | one month
  Number of patients who have taken a counselling session

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospital, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Most probably that IPD can be shared after publication

REFERENCES:
- See also: accessment individual participant data sets and any supporting information is through authorsact cont — https://pubmed.ncbi.nlm.nih.gov/37527416/